CLINICAL TRIAL: NCT00122525
Title: Effect of Safe Male Circumcision on Incidence of Infection by HIV, HSV-2 and of Genital Ulceration
Brief Title: Effect of Male Circumcision on HIV Incidence (ANRS 1265)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: following DSMB recommandation.
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 1265
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: HIV Infections; Herpes Genitalis; Venereal Diseases
Keywords: HIV; Male circumcision; Prevention; HSV-2; Africa; Sexual behavior
MeSH Terms: conditions — HIV Infections; Herpes Genitalis; Sexually Transmitted Diseases; Sexual Behavior | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Male Circumcision

SUMMARY:
Observational studies suggest that male circumcision may provide protection against HIV-1 infection. A randomized, controlled, intervention trial was conducted in a general population of South Africa to test this hypothesis.

DETAILED DESCRIPTION:
This study is a randomized controlled intervention trial. This multi-centre study will take place in 3 centers located around Johannesburg, in the areas of Orange Farm, Sebokeng and Evaton. The intervention group patients (circumcised at the beginning of the trial) and the control group (uncircumcised men) will be followed during 21 months (from M.0 to M. 21). Randomization and medicalized circumcision will be performed at M.0 in the intervention group and might be optional in the control group at end of study. The medicalized circumcision effectiveness will be evaluated on and after M.3 (3 months after medicalized circumcision). Incidences (of HIV, HSV-2 infections and genital ulcer disease) will be compared from M.3 to M.21 between the intervention group and the control group. An intermediate analysis will take place at M. 12.

ELIGIBILITY:
Inclusion Criteria:

* Uncircumcised men aged 18-24 years
* Be in good general condition with normal physical and genital examinations
* Consenting to participate in the trial and to sign an informed consent
* Consenting to randomization of the medicalized circumcision schedule (performed at the beginning of study for the treated group, optional at the end of study for the control group)
* Consenting to avoid sexual contact (except with condom protection) during the 6 weeks following the medicalized circumcision
* Consenting to blood tests at M.0, M.3, M.12 and M.21 tested for HIV, HSV-2 and syphilis.

Exclusion Criteria:

* Men with AIDS
* Men with contraindication for circumcision
* Men thinking of moving away from the trial sites within the 21 months following inclusion
* Men with clinical sexually transmitted diseases (STDs) (those men could be included after treatment)

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3274 (Actual)
Dates: Start 2002-07; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Measure the protective effect of medicalized male circumcision on HIV infection | M3, M12 and M21

SECONDARY OUTCOMES:
Measure the protective effect on infections by the genital herpes agent Herpes simplex virus type 2 (HSV-2) | M3, M12 and M21
Measure the protective effect on the incidence of genital ulcer disease | M3, M12 and M21

CONTACTS AND LOCATIONS:
Overall Officials: Bertran Auvert, MD, Study Chair — Hôpital Ambroise-Paré (AP-HP); Inserm U687; Adrian Puren, Principal Investigator — NICD, Johannesburg, South Africa
Locations (1):
- MC Centre, Orange Farm, Johannesburg, South Africa

REFERENCES:
- [Background] Auvert B, Marseille E, Korenromp EL, Lloyd-Smith J, Sitta R, Taljaard D, Pretorius C, Williams B, Kahn JG. Estimating the resources needed and savings anticipated from roll-out of adult male circumcision in Sub-Saharan Africa. PLoS One. 2008 Aug 6;3(8):e2679. doi: 10.1371/journal.pone.0002679. PMID 18682725
- [Result] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Result] Sobngwi-Tambekou J, Taljaard D, Nieuwoudt M, Lissouba P, Puren A, Auvert B. Male circumcision and Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis: observations after a randomised controlled trial for HIV prevention. Sex Transm Infect. 2009 Apr;85(2):116-20. doi: 10.1136/sti.2008.032334. Epub 2008 Dec 15. PMID 19074928
- [Result] Sobngwi-Tambekou J, Taljaard D, Lissouba P, Zarca K, Puren A, Lagarde E, Auvert B. Effect of HSV-2 serostatus on acquisition of HIV by young men: results of a longitudinal study in Orange Farm, South Africa. J Infect Dis. 2009 Apr 1;199(7):958-64. doi: 10.1086/597208. PMID 19220143
- [Result] Auvert B, Sobngwi-Tambekou J, Cutler E, Nieuwoudt M, Lissouba P, Puren A, Taljaard D. Effect of male circumcision on the prevalence of high-risk human papillomavirus in young men: results of a randomized controlled trial conducted in Orange Farm, South Africa. J Infect Dis. 2009 Jan 1;199(1):14-9. doi: 10.1086/595566. PMID 19086814
- [Derived] Mehta SD, Gray RH, Auvert B, Moses S, Kigozi G, Taljaard D, Puren A, Agot K, Serwadda D, Parker CB, Wawer MJ, Bailey RC. Does sex in the early period after circumcision increase HIV-seroconversion risk? Pooled analysis of adult male circumcision clinical trials. AIDS. 2009 Jul 31;23(12):1557-64. doi: 10.1097/QAD.0b013e32832afe95. PMID 19571722
- See also: Sponsor web page — http://www.anrs.fr